CLINICAL TRIAL: NCT04719065
Title: A Multicenter, Randomized, Open-label, Phase Ib Study to Evaluate the Safety, Efficacy and Pharmacokinetic Characteristics of Mitoxantrone Hydrochloride Liposome Injection in Subjects With Advanced Solid Tumor
Brief Title: A Study of Mitoxantrone Hydrochloride Liposome Injection in the Treatment of Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-017
Record Dates: First submitted 2020-12-14; First posted 2021-01-22 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-08

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A, Mitoxantrone Hydrochloride Liposome Injection, q4w (Experimental): Subjects with advanced or metastatic solid tumor will receive Mitoxantrone Hydrochloride Liposome every 28 days (a cycle) for a maximum of 8 cycles. The starting dose of Mitoxantrone Hydrochloride Liposome is 20mg/m2.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection (IV)
- Group B, Mitoxantrone Hydrochloride Liposome Injection, q3w (Experimental): Subjects with advanced or metastatic solid tumor will receive Mitoxantrone Hydrochloride Liposome every 21 days (a cycle) for a maximum of 8 cycles. The starting dose of Mitoxantrone Hydrochloride Liposome is 20mg/m2.
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection (IV)

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome, intravenous injection (IV) — Subjects will receive Mitoxantrone Hydrochloride Liposome 20 mg/ m2, IV, on day 1 of each cycle for a maximum of 8 cycles.

SUMMARY:
This is a multicenter, randomized, open-label, phase Ib study to evaluate the safety, efficacy and pharmacokinetic characteristics of Mitoxantrone Hydrochloride Liposome in subjects with advanced solid tumor.

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, phase Ib study to evaluate the safety, efficacy and pharmacokinetic characteristics of Mitoxantrone Hydrochloride Liposome in subjects with advanced solid tumor. 90 subjects will be recruited. The first 60 subjects will be randomly assigned into 2 groups, group A and group B. The 30 subjects in group A will receive the Mitoxantrone Hydrochloride Liposome 20 mg/m2 by an intravenous infusion (IV), every 28 days (q4w, 1 cycle). The 30 subjects in group B will receive Mitoxantrone Hydrochloride Liposome 20 mg/m2, IV, every 21 days (q3w, 1 cycle). After this, the last 30 subjects will be assigned into group B. All subjects will receive the treatment until disease progression, intolerable toxic reaction, death, or withdrawal by investigator or subject decision (a maximum of 8 cycles). Delays in drug administration is allowed from cycle 2, however, the delays should be no more than 3 weeks. Dose adjustments after cycle 2 is permitted, and the minimum dose is 12 mg/m2.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent;
2. Age ≥18, without gender limitation;
3. Histologically and/or cytologically confirmed diagnosis of unresectable local or metastasizing advanced solid tumor;
4. Fail to respond to standard therapy or lack of effective treatment, including no standard therapy, intolerance of standard therapy, etc.;
5. At least one measurable lesion according to RECIST v1.1;
6. ECOG performance status of 0 or 1;
7. AEs from the previous treatment have resolved to ≤ Grade 1 based on CTCAE (except for the toxicity without safety risk judged by the investigator, such as hair loss, hyperpigmentation);
8. Adequate organ function;
9. Subjects of childbearing potential must agree to use effective contraceptive measures. Female subjects must have a negative pregnancy test before enrollment;
10. Fully comply with the protocol.

Exclusion Criteria:

1. History of allergy to mitoxantrone hydrochloride or any excipients of the study drug;
2. Untreated or symptomatic central nervous system (CNS) metastases;
3. CTCAE Grade 3 or Grade 4 gastrointestinal hemorrhage within 12 weeks prior to the first dose administration;
4. History of allotransplantation;
5. Known hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or other active viral infection;
6. Serious infection or interstitial pneumonia within 1 week prior to the first dose administration;
7. Use of other anticancer treatment within 4 weeks prior to the first dose administration;
8. Enrolled in any other clinical trials within 4 weeks prior to the first dose administration;
9. Major surgery within 3 months prior to the first dose administration, or have a surgical schedule during the study period;
10. Thrombosis or thromboembolism within 6 months prior to screening;
11. History of, or known additional malignant tumor within 3 years, except for tumors have been cured and have not recurred, and carcinoma in situ;
12. Impaired cardiac function or serious cardiac disease;
13. Previous treatment with adriamycin or other anthracyclines, and the total cumulative dose of prior adriamycin or equivalent is >350 mg/m2;
14. Life expectancy<12 weeks;
15. Pregnant or lactating female;
16. Serious and/or uncontrolled systemic diseases;
17. Not suitable for this study as decided by the investigator due to other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-13 (Actual); Primary Completion 2022-04-13 (Estimated); Study Completion 2024-04-13 (Estimated)

PRIMARY OUTCOMES:
adverse events (AEs) | from the first dose injection to 28 days after the last dose injection, assessed up to 36 weeks
  The incidence and severity of AEs, abnormalities in physical exams, vital sign assessments, clinical laboratory assessments, ultrasonic cardiograms (UCGs) and electrocardiographs (ECGs).

SECONDARY OUTCOMES:
overall response rate (ORR) | From the enrollment to the final documentation of response of the last subject (assessed up to 36 months)
  To investigate the preliminary antitumor efficacy
duration of response (DoR) | From the enrollment to CR,PR, PD, death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy
duration of complete response (DCR) | From the enrollment to the final documentation of response of the last subject (assessed up to 36 months)
  To investigate the preliminary antitumor efficacy
progression-free survival (PFS) | From the enrollment to CR,PR, PD, death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy
overall survival (OS) | From the enrollment to CR, PR, PD, death, lost to follow-up, withdrawal, or study end, whichever occurred first, assessed up to 36 months
  To investigate the preliminary antitumor efficacy
maximum time (Tmax) | Cycle 1 to cycle 4, approximately 16 weeks
  To investigate PK characteristics
maximum concentration (Cmax) | Cycle 1 to cycle 4, approximately 16 weeks
  To investigate PK characteristics
area under the plasma concentration-time curve from time zero to the time of last observed concentration (AUC0-t) | Cycle 1 to cycle 4, approximately 16 weeks
  To investigate PK characteristics
apparent terminal half-life (t1/2) | Cycle 1 to cycle 4, approximately 16 weeks
  To investigate PK characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Yehui Shi, MD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (8):
- China (8):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No